CLINICAL TRIAL: NCT03929640
Title: Management Of Pain After Cesarean Trial
Acronym: MOPAC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lead co-I left institution in 2020 and enrollment was suspended. Study was kept open in hopes of finding a replacement/meeting enrollment goal, but a new lead was not found. Study is now officially closed.
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Serdar Ural, Professor, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00010393
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ibuprofen and placebo (Placebo Comparator): Oral administration of ibuprofen 600 mg tablet and placebo tablet every 6 hours
  Interventions: Drug: Placebo; Drug: Ibuprofen
- Ibuprofen and acetaminophen (Active Comparator): Oral administration of ibuprofen 600 mg tablet and acetaminophen 650 mg tablet every 6 hours
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen 650 mg tablet every 6 hours
  Arms: Ibuprofen and acetaminophen
Drug: Placebo — Placebo oral tablet every 6 hours
  Arms: Ibuprofen and placebo
Drug: Ibuprofen — Ibuprofen 600 mg tablet every 6 hours

SUMMARY:
This is a double blinded randomized controlled trial to test the efficacy of a combination of acetaminophen and ibuprofen administered to patients on schedule compared to ibuprofen alone on the patient's reported pain score on the second post-operative day after Cesarean delivery. The investigators will also record opiate consumption and pain scores throughout the hospitalization of participants, and will survey patients at one and two weeks after surgery regarding opiate consumption and quality of life.

DETAILED DESCRIPTION:
The investigators have designed a double-blinded randomized, controlled trial to compare a standardized pain regimen of scheduled ibuprofen and acetaminophen to scheduled ibuprofen and placebo. In both arms, the participant will have the ability to ask for medication for breakthrough pain which will be oxycodone. By standardizing and scheduling the administration of ibuprofen with acetaminophen, the investigators hypothesize that total opioid requested and therefore consumed will be decreased in this participants who receive ibuprofen scheduled with acetaminophen. The investigators will primarily assess pain as reported on a 10-point scale mid-day on the second post-operative day. Secondarily, the investigators will collect reported pain scores and total opiate consumption while in the hospital, opiate consumption after discharge, and quality of life as assessed by the World Health Organization Quality of Life "Bref" (WHOQOL-BREF) survey. This information will be obtained via chart review and at-home surveys administered via email on the Research Electronic Data Capture (REDCap) system one and two weeks after surgery.

Enrollment will be performed by study staff. Participants will then be randomized by the institution's Investigational Drug Services (IDS) in REDCap, which uses a randomization table generated by Penn State University (PSU) bio-statisticians. A medication packet will then be prepared and distributed by IDS for the participant containing 20 tablets of acetaminophen 650 mg or placebo based on randomization assignment. The packet will then be sent to nursing staff caring for the patient. Participants will then receive study medication/placebo along with ibuprofen 600 mg (dispensed by the clinical pharmacy) every 6 hours. Participants will be able to request medication for breakthrough pain which will be oxycodone 5 mg or 10 mg depending on reported pain score (one pill for moderate pain, two pills for severe pain). Both ibuprofen and oxycodone will be ordered and dispensed by the clinical pharmacy. Until the participant is deemed able to receive medication by mouth, the participant may receive medication as prescribed by the caring obstetrician and/or anesthesiologist which will be beyond the scope of this trial. Pain scores will be collected and recorded in the medical chart by nursing and assistant staff as part of routine care.

At discharge, participants will receive a standard prescription for 20 tablets of oxycodone 5 mg with directions to take 1-2 tablets every 6-8 hours as needed for breakthrough pain, as is the current group standard at the institution in the Department of Obstetrics and Gynecology.

After discharge, study staff will then conduct a chart review to collect demographic information, review the operative report, and ensure no event took place which would exclude the participant from the study. Study staff will also record total opiate consumption and pain scores.

One week after surgery, the participant will receive an invitation via electronic mail (e-mail) to complete a survey on REDCap which will assess opiate consumption and perceived appropriateness of pain control. Two weeks after surgery, participants will receive two additional invitations; one to complete another survey to assess opiate consumption and perceived appropriateness of pain control, and a second to complete the WHOQOL-BREF. The WHOQOL-BREF survey has been validated to assess four distinct categories of quality of life in women two weeks postpartum. These invitations and reminders have been designed to occur automatically with the assistance of features inherent to the REDCap program. Participants will be considered non-compliant if they fail to complete surveys within three days of receiving their invitation.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at least 18 years of age
* Planned delivery via C-section
* Pfannenstiel skin incision
* Lower uterine segment transverse hysterotomy
* English speaking

Exclusion Criteria:

* Major intra-operative or post-operative complication such that clinician recommends patient should not receive non-steroidal anti-inflammatory drugs or that patient requires acetaminophen to treat fever (ie suspected endometritis)
* Unplanned surgery (hysterectomy, bowel/bladder repair)
* Allergy or contraindication to study medication
* Non-English speaking
* Inability to provide informed consent
* History of opioid, other illicit substance, or alcohol use disorder either before or during pregnancy
* Severe renal or hepatic impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women may participate due to pregnancy-related condition being studied
Enrollment: 49 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-03-14 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pennsylvania State University Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
May collaborate with PSU Addiction Center to perform secondary analyses on data collected, including total opiate consumption and pain scores.

REFERENCES:
- [Background] Bateman BT, Cole NM, Maeda A, Burns SM, Houle TT, Huybrechts KF, Clancy CR, Hopp SB, Ecker JL, Ende H, Grewe K, Raposo Corradini B, Schoenfeld RE, Sankar K, Day LJ, Harris L, Booth JL, Flood P, Bauer ME, Tsen LC, Landau R, Leffert LR. Patterns of Opioid Prescription and Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):29-35. doi: 10.1097/AOG.0000000000002093. PMID 28594763
- [Background] Bartels K, Mayes LM, Dingmann C, Bullard KJ, Hopfer CJ, Binswanger IA. Opioid Use and Storage Patterns by Patients after Hospital Discharge following Surgery. PLoS One. 2016 Jan 29;11(1):e0147972. doi: 10.1371/journal.pone.0147972. eCollection 2016. PMID 26824844
- [Background] Osmundson SS, Schornack LA, Grasch JL, Zuckerwise LC, Young JL, Richardson MG. Postdischarge Opioid Use After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):36-41. doi: 10.1097/AOG.0000000000002095. PMID 28594766
- [Background] Prabhu M, McQuaid-Hanson E, Hopp S, Burns SM, Leffert LR, Landau R, Lauffenburger JC, Choudhry NK, Kaimal A, Bateman BT. A Shared Decision-Making Intervention to Guide Opioid Prescribing After Cesarean Delivery. Obstet Gynecol. 2017 Jul;130(1):42-46. doi: 10.1097/AOG.0000000000002094. PMID 28594762
- [Background] Viteri OA, England JA, Alrais MA, Lash KA, Villegas MI, Ashimi Balogun OA, Chauhan SP, Sibai BM. Association of Nonsteroidal Antiinflammatory Drugs and Postpartum Hypertension in Women With Preeclampsia With Severe Features. Obstet Gynecol. 2017 Oct;130(4):830-835. doi: 10.1097/AOG.0000000000002247. PMID 28885417
- [Background] Chang AK, Bijur PE, Esses D, Barnaby DP, Baer J. Effect of a Single Dose of Oral Opioid and Nonopioid Analgesics on Acute Extremity Pain in the Emergency Department: A Randomized Clinical Trial. JAMA. 2017 Nov 7;318(17):1661-1667. doi: 10.1001/jama.2017.16190. PMID 29114833
- [Background] Ong CK, Seymour RA, Lirk P, Merry AF. Combining paracetamol (acetaminophen) with nonsteroidal antiinflammatory drugs: a qualitative systematic review of analgesic efficacy for acute postoperative pain. Anesth Analg. 2010 Apr 1;110(4):1170-9. doi: 10.1213/ANE.0b013e3181cf9281. Epub 2010 Feb 8. PMID 20142348
- [Background] Skevington SM, Lotfy M, O'Connell KA; WHOQOL Group. The World Health Organization's WHOQOL-BREF quality of life assessment: psychometric properties and results of the international field trial. A report from the WHOQOL group. Qual Life Res. 2004 Mar;13(2):299-310. doi: 10.1023/B:QURE.0000018486.91360.00. PMID 15085902

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
Started (Randomized subjects) | 24 | 25
Received Study Drug (Met final eligibility criteria/received study drug) | 20 | 21
Completed (Completed 2w survey) | 18 | 16
Not Completed | 6 | 9

BASELINE CHARACTERISTICS:
Population: Eligible subjects who received study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen | Total
Number analyzed (Participants) | 20 | 21 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.6 (5.0) | 30.0 (9.8) | 30.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 21 | 41
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 7 | 10
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 14 | 12 | 26
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain score on a scale of 0 (no pain) to 10 (worst pain); "pain score" is a verbal report of participant pain on a scale of 0-10, 0 indicating no pain and incrementally increasing as integer to a maximum score of 10 indicating the most severe pain possible.
Time Frame: Post-operative day 2, corresponding to 2 days after cesarean section surgery (day of surgery is considered post-operative day 0). Measurement taken mid-day (12 PM - 4 PM)
Population: Participants having a post-op day 2 (mid-day) pain score in their charts.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
Number analyzed (Participants) | 17 | 17
score on a scale | 3.5 (2.3) | 3.3 (2.4)

2. Secondary Outcome: Opiate Consumption in Hospital
Description: Total number of oxycodone 5 mg tablets taken during hospital admission after cesarean section surgery
Time Frame: Post-operative day 0 (day of surgery) until discharged from hospital on post-operative day 3 or 4.
Population: Subjects with available data in their charts
Measure: Median (Inter-Quartile Range); unit: number of tablets
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
Number analyzed (Participants) | 18 | 20
number of tablets | 10 [1 to 20] | 9 [0 to 17]

3. Secondary Outcome: WHOQOL-BREF Score, Domain 1
Description: Domain Score on World Health Organization Quality of Life - Brief (WHOQOL-BREF) survey. The survey consists of 26 questions and evaluates four domains of quality of life including physical health (domain 1), psychological (domain 2), social relationships (domain 3), and environment (domain 4). Domain scores are scaled in a positive direction (i.e. higher scores denote higher quality of life) and range between 4-20, comparable with the WHOQOL-100.
Time Frame: Post-operative Day 14 (two weeks after cesarean section surgery)
Population: subjects completing this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
Number analyzed (Participants) | 16 | 18
score on a scale | 15.6 (2.3) | 16.2 (2.6)

4. Secondary Outcome: WHOQOL-BREF Score, Domain 2
Description: as for outcome 3
Time Frame: Post-operative Day 14 (two weeks after cesarean section surgery)
Population: subjects completing this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
Number analyzed (Participants) | 16 | 18
score on a scale | 15.6 (2.8) | 16.4 (1.7)

5. Secondary Outcome: WHOQOL-BREF Score, Domain 3
Description: as for outcome 3
Time Frame: Post-operative Day 14 (two weeks after cesarean section surgery)
Population: subjects completing this survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
Number analyzed (Participants) | 16 | 18
score on a scale | 15.4 (2.9) | 17.1 (2.3)

6. Secondary Outcome: WHOQOL-BREF Score, Domain 4
Description: as for outcome 3
Time Frame: Post-operative Day 14 (two weeks after cesarean section surgery)
Population: subjects who completed the survey
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
Number analyzed (Participants) | 16 | 18
score on a scale | 17.2 (1.8) | 17.1 (1.6)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Ibuprofen and Placebo | Ibuprofen and Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/21
Other Adverse Events (participants affected / at risk) | 0/20 | 0/21

LIMITATIONS AND CAVEATS:
Enrollment was suspended when the co-investigator responsible for study recruitment left the institution in 2020. At that time, only 49 subjects had been randomized (study enrollment goal was 150 subjects). The PI kept the study open but was not successful in finding a replacement to lead the study so it was eventually terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03929640/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-20): https://cdn.clinicaltrials.gov/large-docs/40/NCT03929640/ICF_001.pdf